CLINICAL TRIAL: NCT05191329
Title: Impact of Personality Type, Social Roles and Working Mandates οn Visual Capacity and Satisfaction of Patients That Underwent Pseudophakic Presbyopic Correction
Brief Title: Impact of Personality on Satisfaction Following Presbyopic Correction
Status: Completed | Type: Observational
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Georgios Labiris, Associate Professor, Democritus University of Thrace
Other Study IDs: 844/18-09-2018
Record Dates: First submitted 2021-12-30; First posted 2022-01-13 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Personality; Patient Satisfaction; Presbyopia
Keywords: multifocal presbyopic correction; personality traits; vision oriented quality of life
MeSH Terms: conditions — Patient Satisfaction; Presbyopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: 40 patients with non surgical presbyopic correction e.g. glasses and 80 patients that underwent pseudophakic presbyopic correction with multifocal or trifocal IOLs
  Interventions: Diagnostic Test: TPQue Greek version, NEI-VFQ-25 Greek version

INTERVENTIONS:
Diagnostic Test: TPQue Greek version, NEI-VFQ-25 Greek version — Study participants with non surgical presbyopic correction will be evaluated with TPQue regarding their personality traits. Visual acuity will also be assessed. Study participants with pseudophakic presbyopic correction will be evaluated with the TPQue before surgery. They will also be visual acuity evaluation and NEI-VFQ-25 assessment six months after surgery.

SUMMARY:
Primary objective of this study is the exploration of the impact of personality type, social roles and working mandates οn the visual capacity and satisfaction of patients that underwent pseudophakic presbyopic correction.

DETAILED DESCRIPTION:
Personality type, social types and working mandates will be evaluated as a routine procedure to patients that visit the Presbyopia Service of the University Hospital of Alexandroupolis, by means of structured questionnaires. Six months following pseudophakic presbyopic correction surgery, each study participant will be evaluated for his/her visual capacity and vision-specific quality of life. Regression modeling will be attempted in order to identify the exact demographics, social roles and personality type of the patient that is most compatible to receive pseudophakic presbyopic correction.

ELIGIBILITY:
Inclusion Criteria:

* presbyopia, patients of our outpatient ophthalmology clinic, age between 40 and 85 years

Exclusion Criteria:

* inability to cooperate, former diagnosis of mental disease

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: participants with presbyopia, either surgically or non surgically corrected, aged 40 to 85 years
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-08-28 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
TPQue assessment | 6 months
  Participants' personality traits will be evaluated by the examiner using the Greek version of the Traits Personality (TPQue) questionnaire, with a scale from 0 to 100. 100 is the highest percentage of a certain trait.
NEI-VFQ-25 assessment | 6 months
  Participants' vision oriented quality of life will be assessed using the Greek version of the National Eye Institute Visual Function Questionnaire-25 (NEI VFQ-25), with a scale from 0 to 100. 100 being the highest satisfaction rate.

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Labiris, MD,PhD, Study Chair — Department of Ophthalmology, University Hospital of Alexandroupolis, Alexandroupolis, Greece
Locations (1):
- Department of Ophthalmology, University Hospital of Alexandroupolis, Alexandroupoli, Evros, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ntonti P, Bakirtzis M, Delibasis K, Seimenis I, Tsinopoulos I, Labiris G. Impact of personality on the decision process and on satisfaction rates in pseudophakic presbyopic correction. J Cataract Refract Surg. 2022 Dec 1;48(12):1433-1439. doi: 10.1097/j.jcrs.0000000000001021. PMID 35862830